CLINICAL TRIAL: NCT01459419
Title: A Phase IIa Safety Study of Oral Administration of Anti-CD3 Monoclonal Antibody in Non-responder Genotype-I Chronic Hepatitis C Subjects, a Single-blind, Randomized, Controlled Multi-center Study.
Brief Title: Oral Administration of Anti-CD3 Monoclonal Antibody in Non-responder Genotype-I Chronic Hepatitis C Subjects
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Inspira Medical AB (Industry)
Collaborators: NasVax Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ISM-10-06
Record Dates: First submitted 2011-10-23; First posted 2011-10-25 (Estimated); Last update posted 2011-10-25 (Estimated); Status verified 2011-10

CONDITIONS: Chronic Hepatitis C
MeSH Terms: conditions — Hepatitis C, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- anti-CD3 monoclonal antibody (Experimental): Oral anti-CD3 MAb will be administered at a dosage level of 0.2 or 1.0 or 5.0 mg per day for 30 days. Up to 9 subjects will be treated at each dosage level
  Interventions: Drug: anti-CD3 monoclonal antibody
- Sodium chloride (Placebo Comparator): Up to 9 subjects will receive placebo. Subjects will receive the drug in a similar manner as as the treatment group
  Interventions: Drug: Sodium Chloride placebo

INTERVENTIONS:
Drug: anti-CD3 monoclonal antibody — Oral anti-CD3 MAb will be administered at a dosage level of 0.2 or 1.0 or 5.0 mg per day for 30 days. One 20mg tablet of Omeprazole (a proton pump inhibitor) will be taken concomitantly orally
  Arms: anti-CD3 monoclonal antibody
Drug: Sodium Chloride placebo — Sodium chloride will be administered orally every day for 30 days. Up to 9 subjects will be treated at each dosage level. One 20mg tablet of Omeprazole (a proton pump inhibitor) will be taken concomitantly orally
  Arms: Sodium chloride

SUMMARY:
The use of oral aCD3 Monoclonal antibody (MAb) alone in subjects with hepatitis C is justified on the basis of scientific and medical reasons. There are data in multiple animal models that aCD3-alone confers efficacy in models of inflammatory or autoimmune disease and induces regulatory T cells and immune-modulation as desired in clinical studies. These observations are reinforced by data in the Phase 1 clinical study showing that aCD3-alone induced the desired immune-modulation in terms of immunological markers for regulatory T cells and appropriate rises and declines in certain cytokine levels.

DETAILED DESCRIPTION:
Oral aCD3 MAb will be administered at a dosage level of 0.2 or 1.0 or 5.0 mg per day for 30 days. Up of 9 subjects will be treated at each dosage level, and up to 9 subjects will receive placebo buffered in normal saline that is used as diluents for the MAb. One 20mg tablet of Omeprazole (a proton pump inhibitor) will be taken orally as part of the study drug cocktail in order to neutralize stomach pH for enhancing stability of the MAb. During the treatment period, subjects will ingest the study drug/s every day for 30 days, and will be followed for clinical and laboratory effects. Subjects will be followed up to Day 60 (30 days after termination of treatment)

ELIGIBILITY:
* Subjects who have completed the informed consent process culminating with written informed consent by the subject.
* Men and women age 18 to 65 years (inclusive).
* Diagnosis of chronic active HCV infection was based on liver biopsy (within 3 years of initiation of study),
* Patients who failed treatment with Interferon or Peg-Interferon and Ribavirin (<2-log change in HCV level during the 12 weeks of treatment)
* HCV RNA in blood for at Screening Visit, ≥600 copies/mL
* Abstinence from any alternative medications or vitamin-D-containing supplements for three months prior to initiation of therapy was stipulated.
* Compensated liver disease with the following maximum hematologic, biochemical and serologic criteria at the Screening visit (WNL=within normal limits) Hemoglobin ≥ 12 g/dl for women and ≥ 13 g/dl for men, WBC > 3000/mm3, Platelets > 100,000/mm3, Direct bilirubin - WNL. Indirect bilirubin - WNL, Albumin - WNL, Serum Creatinine - WNL. Child-Pugh score ≤ 6.
* Fasting glucose should be 70 -140 mg/dl, results between 116-140 require HbA1c < 7.5%
* Antinuclear antibodies (ANA) up to +1
* HCV Genotype I patients

Exclusion Criteria:

* Subjects who have undergone surgery within the last 3 months.
* Subjects who have had a prior gastrointestinal surgery.
* Subjects with organ transplants other than cornea or hair transplant.
* Subjects with Inflammatory Bowel Disease, malabsorption, and symptoms of diarrhea.
* Subjects with a clinically significant (during last 3 months) infectious, immune-mediated or malignant disease.
* Subjects who are receiving an elemental diet or parenteral nutrition.
* Subjects who have been treated with any type of immune modulatory drug including systemic steroids or NSAID within the last 4 weeks.
* Subjects who have received either methotrexate or cyclosporine or anti-TNF (infliximab, Remicade) or anti-integrin (namixilab) at any time or who have participated in any other clinical trial within the last 3 months.
* Subjects with a history of coagulopathy.
* ALT level more than 10 times the normal limit.
* Women with childbearing potential unless using adequate contraception (either IUD, oral or Depo-provera contraceptive, or barrier plus spermicide); pregnant or breastfeeding mothers.
* Subjects who will be unavailable for the duration of the trial, who are unlikely to be compliant with the protocol, or who are felt to be unsuitable by the Investigator for any other reason.
* Subjects who are HIV-positive.
* Subjects who are positive for anti-HBcAg
* Subjects with active CMV infection.
* Subjects with autoimmune hepatitis
* Subjects with IgG anti-cardiolipin antibody >16 IU.
* Any prior exposure to anti-CD3 MAb.
* Known sensitivity to any ingredients in the study drug
* Any know autoimmune disease except for the studied disorders
* Subjects with excess alcohol use (> 30 g/day)
* Subjects with drug addiction based on the physician's judgment
* Subjects with TSH >6 mIU/L

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2011-11; Primary Completion 2013-05 (Estimated); Study Completion 2013-10 (Estimated)

PRIMARY OUTCOMES:
This clinical study is designed to evaluate as Primary Objective the safety of oral administration of the study drug anti-CD3 MAb to non responder genotype I subjects with the chronic Hepatitis C. | 60
  The safety and tolerability of oral administration of the study drug cocktail will be evaluated at Days 7, 14, 21 and 30 by physical examinations and thorough medical history and laboratory evaluations as described below and by the subject through his/her diary entries. In addition, subjects will be assessed for safety at Day 60

SECONDARY OUTCOMES:
Decrease in the concentration of HCV | 30 days
  30 days
Liver function test | 30 days
  Changes in ALT will be used to evaluate effect on liver

CONTACTS AND LOCATIONS:
Overall Officials: Waldemar Halota, Prof, Principal Investigator — Katedra i Klinika Chorób Zakaźnych i Hepatologii Wojewódzki Szpital Obserwacyjno - Zakaźny im. Tadeusza Browicza
Locations (2):
- Univ.Klinik für Innere Medizin IV, Vienna, Austria
- Katedra i Klinika Chorób Zakaźnych i Hepatologii Wojewódzki Szpital Obserwacyjno - Zakaźny im. Tadeusza Browicza, Bydgoszcz, Bydgoszcz, Poland